CLINICAL TRIAL: NCT02546336
Title: Ultrasound-Guided Hip Joint Cooled Radiofrequency Denervation: A Prospective Pilot Study
Brief Title: Ultrasound-Guided Hip Joint Cooled Radiofrequency Denervation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staff for the study is no longer available.
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIP RFD
Record Dates: First submitted 2015-08-13; First posted 2015-09-10 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hip Osteoarthritis; Chronic Pain
Keywords: Ultrasound Guidance; Cooled Radiofrequency; Hip Denervation
MeSH Terms: conditions — Osteoarthritis, Hip; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-Guided Hip Denervation (Experimental): This is a pilot study. 15 Hip Osteoarthritis patients with chronic pain will be recruited in this pilot arm. These will undergo Ultrasound-Guided Cooled Radiofrequency Hip Denervation as intervention.
  Interventions: Device: Ultrasound-Guided Cooled Radiofrequency Hip Denervation

INTERVENTIONS:
Device: Ultrasound-Guided Cooled Radiofrequency Hip Denervation — Light neuroleptic anesthesia and skin preparation will be performed. Under Ultrasound guidance, an active probe will be inserted. Sensory and motor stimulation will be administered. Anteroposterior fluoroscopy image will be recorded. Lesioning of articular branches of femoral and obturator nerves via radiofrequency will be performed after lidocaine injection. WOMAC, EQ-5D and SF-12 questionnaires will be used for measuring outcomes postoperatively.

SUMMARY:
Hip osteoarthritis (HOA) is a common cause of pain and disability in aging population. Conservative treatment is based on lifestyle modifications, physical therapy, analgesic and anti-inflammatory medications and intra articular injections. This Prospective Pilot Study aims at investigating the efficacy of Ultrasound-Guided Cooled Radiofrequency Hip Denervation as a treatment offered to patients with HOA.

DETAILED DESCRIPTION:
Radiological prevalence of HOA is very high. Hip denervation (HD) is a known palliative procedure that was initially performed as an open surgery. The role of the obturator, femoral and sciatic nerves in hip joint innervation was discovered. Several small clinical and anatomical studies addressed feasibility and benefits of the radiofrequency hip denervation (RFHD). Ultrasound guidance may eliminate equivocality of previously published techniques and provide precise image guidance as it a is logical and anatomically sound approach when procedural targets include soft tissue, such as nerves, tendons and joint capsule. None of these structures can be localized under routine fluoroscopy. Ultrasound is a bedside imaging tool that has been accepted as safe and reliable. In two meta-analyses, the use of real-time two-dimensional ultrasound for the placement of CVCs substantially decreased mechanical complications and reduced the number of attempts at required cannulation and failed attempts at cannulation compared with the standard landmark placement. Pertinent to the proposed study, recent systematic review and meta-analysis of the accuracy of US-guided versus landmark-guided hip joint injections revealed that US-guided injections are significantly more accurate than those that are landmark-guided. The significance of this study lies in its potential to improve functional activity and pain control in patients with HOA. Also, it may eventually lead to a decrease in patients resorting to Total Hip Arthroplasty (THA) as an ultimate end solution for HOA.

ELIGIBILITY:
Inclusion Criteria:

* Primary degenerative osteoarthritis of hip joint
* Pain pre-intervention qualified as at least moderate with functional limitation moderate/severe.
* Radiological confirmation of hip osteoarthritis
* Failure of conservative therapy to control symptoms, defined as the persistence of at least moderate with functional limitation moderate/severe pain that has been refractory to prescribed medications, and other modalities, such as physical therapy and intraarticular injections. Intolerable side effects of medications and contraindications to specific methods will be also considered as a failure of the conservative therapy.
* Positive articular branches analgesic block, defined as >50% improvement in pain and function for at least 2 hours

Exclusion Criteria:

* Non-English speakers
* Daily dose of opioids more than 90 MEQ
* Body Mass Index (BMI) > 30
* Uncorrectable coagulopathy
* Local and systemic infection
* Inability to obtain ultrasound image of ventral acetabulum
* Documented prior Anaphylactic Reaction to Contrast Agent
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario and MacMaster Universities Osteoarthritis Index (WOMAC) Score | 12 months
  A questionnaire designed to assess pain, stiffness, and physical function in patients with hip and/or knee osteoarthritis (OA)1
  The WOMAC consists of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing Stiffness (2 items): after first waking and later in the day Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.

SECONDARY OUTCOMES:
Short Form (12) Health Survey (SF-12) | 12 months
  A generic, multipurpose short-form survey with 12 questions selected from the SF-36 Health Survey which, when combined, scored and weighted, results in two scales of mental and physical functioning and overall health-related quality of life.
EQ-5D | 12 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It is applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. It is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gofeld, MD, FIPP, Principal Investigator — Women's College Hospital/ Saint Michael's Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Nelson AE, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of hip symptoms and radiographic and symptomatic hip osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2009 Apr;36(4):809-15. doi: 10.3899/jrheum.080677. Epub 2009 Mar 13. PMID 19286855
- [Background] Vincent HK, Heywood K, Connelly J, Hurley RW. Obesity and weight loss in the treatment and prevention of osteoarthritis. PM R. 2012 May;4(5 Suppl):S59-67. doi: 10.1016/j.pmrj.2012.01.005. PMID 22632704
- [Background] Brakke R, Singh J, Sullivan W. Physical therapy in persons with osteoarthritis. PM R. 2012 May;4(5 Suppl):S53-8. doi: 10.1016/j.pmrj.2012.02.017. PMID 22632703
- [Background] MULDER JD. Denervation of the hip joint in osteoarthritis. J Bone Joint Surg Br. 1948 Aug;30B(3):446-8. No abstract available. PMID 18877978
- [Background] Akatov OV, Dreval ON. Percutaneous radiofrequency destruction of the obturator nerve for treatment of pain caused by coxarthrosis. Stereotact Funct Neurosurg. 1997;69(1-4 Pt 2):278-80. doi: 10.1159/000099888. PMID 9711767
- [Background] Rivera F, Mariconda C, Annaratone G. Percutaneous radiofrequency denervation in patients with contraindications for total hip arthroplasty. Orthopedics. 2012 Mar 7;35(3):e302-5. doi: 10.3928/01477447-20120222-19. PMID 22385437
- [Background] Kawaguchi M, Hashizume K, Iwata T, Furuya H. Percutaneous radiofrequency lesioning of sensory branches of the obturator and femoral nerves for the treatment of hip joint pain. Reg Anesth Pain Med. 2001 Nov-Dec;26(6):576-81. doi: 10.1053/rapm.2001.26679. PMID 11707799
- [Background] Malik A, Simopolous T, Elkersh M, Aner M, Bajwa ZH. Percutaneous radiofrequency lesioning of sensory branches of the obturator and femoral nerves for the treatment of non-operable hip pain. Pain Physician. 2003 Oct;6(4):499-502. PMID 16871303
- [Background] Fukui S, Nosaka S. Successful relief of hip joint pain by percutaneous radiofrequency nerve thermocoagulation in a patient with contraindications for hip arthroplasty. J Anesth. 2001;15(3):173-5. doi: 10.1007/s005400170023. No abstract available. PMID 14566519
- [Background] Hoeber S, Aly AR, Ashworth N, Rajasekaran S. Ultrasound-guided hip joint injections are more accurate than landmark-guided injections: a systematic review and meta-analysis. Br J Sports Med. 2016 Apr;50(7):392-6. doi: 10.1136/bjsports-2014-094570. Epub 2015 Jun 10. PMID 26062955
- [Background] Gupta G, Radhakrishna M, Etheridge P, Besemann M, Finlayson RJ. Radiofrequency denervation of the hip joint for pain management: case report and literature review. US Army Med Dep J. 2014 Apr-Jun:41-51. PMID 24706242
- [Background] Chaiban G, Paradis T, Atallah J. Use of ultrasound and fluoroscopy guidance in percutaneous radiofrequency lesioning of the sensory branches of the femoral and obturator nerves. Pain Pract. 2014 Apr;14(4):343-5. doi: 10.1111/papr.12069. Epub 2013 May 9. PMID 23656575